CLINICAL TRIAL: NCT00965614
Title: To Validate the Specific Patterns of Magnetocardiography, a Non-invasive Non-contact Examination for Patients With Ischemic Heart Disease or Cardiac Arrhythmia
Status: Available | Type: Expanded Access
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 34MD01
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Arrhythmia
Keywords: diagnose cardiac arrhythmia and CAD.; we'll try to establish the specific model to detect and diagnose cardiac arrhythmia and CAD.
MeSH Terms: conditions — Arrhythmias, Cardiac

INTERVENTIONS:
Other: MCG — Cardiac Arrhythmia,Heart Disease

SUMMARY:
ECG is one of the most important non-invasive method to diagnose CAD and arrhythmia. However, clinically it still has its limitation. Because the electrical field could induce a magnetic field, the newly developed non-contact technique, magnetocardiography, was established to detect the local magnetic field component of the heart. It is safe and more convenient. In this study, we try to define and validate the magnetocardiographic patterns in the patients with cardiac arrhythmias or ischemia.

ELIGIBILITY:
Patient enrollment:

* patients older than 18 years old,
* having received 1) 12-lead ECG examination for suspected cardiac arrhythmias or 2) stress tests for suspected coronary artery disease, will be invited.
* The patients who have medical devices made of metallic or magnetic material (ex. pacemaker, mechanical valve and arthroplasty) will be excluded to prevent the experimental bias.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult